NCT # NCT03107611

**Study Identification Code** CD-14-875

**Statistical Analysis Plan** 

Version 1.0

**Issue Date** June 29, 2017

Study Title A Randomized, Prospective, Multicenter, Double Blind,

Parallel Assignment, Placebo Controlled Bioequivalence

Study of Pimecrolimus Cream, 1% and Elidel® (Pimecrolimus) Cream, 1% in Patients with Mild to

Moderate Atopic Dermatitis

**Sponsor** DPT Laboratories, Ltd., an affiliate of Mylan Inc.

#### **DPT** Laboratories

# Protocol No. CD-14-875 Novella Study No. CT991616

# A RANDOMIZED, PROSPECTIVE, MULTICENTER, DOUBLE BLIND, PARALLEL ASSIGNMENT, PLACEBO CONTROLLED BIOEQUIVALENCE STUDY OF PIMECROLIMUS CREAM, 1% AND ELIDEL® (PIMECROLIMUS) CREAM, 1% IN PATIENTS WITH MILD TO MODERATE ATOPIC DERMATITIS

# Statistical Analysis Plan

**June 29, 2017** 

Novella Clinical (formerly TKL Research Clinical Trials Division)
365 West Passaic Street
Rochelle Park, NJ 07662

Version 1.0 Revision History:

Kathleen Ocasio Director, Clinical Programs DPT Laboratories

Katrin Beckmann Senior Statistician Mylan Healthcare GmbH

Carol Udell, MS
Senior Director, Data Management and
Biostatistics
Novella Clinical

DocuSigned by: 07-Jul-2017 | 06:38:00 PDT Signature Signer Name: Kathleen Ocasio Date Signing Reason: I approve this document Signing Time: 7/7/2017 6:37:52 AM PDT Docusioned by FFE08E0FE0E3411F89EFD4D82881E0930-Jun-2017 | 02:15:07 PDT Signature Signer Name: Katrin Beckmann Date Signing Reason: I approve this document Signing Time: 6/30/2017 2:14:26 AM PDT Preventation | 07:56:42 PDT Date Signature Carol Udell Signing Reason: I approve this document Signing Time: 6/29/2017 7:56:38 AM PDT CE741CD0FE9741ECA29CB39E84B183BB

# **Table of Contents**

| Tab | ole of Contents | 2 |
|-----|-----------------------------------------------|----|
| 1. | INTRODUCTION | 5 |
| 2. | STUDY OBJECTIVES | 5 |
| 3. | STUDY DESIGN | 5 |
| 4. | HARDWARE AND SOFTWARE | 6 |
| 5. | DATABASE CLOSURE | 7 |
| 6. | SAMPLE SIZE DETERMINATION | 7 |
| 7. | HANDLING OF DROPOUTS AND MISSING DATA | 7 |
| 8. | ANALYSIS POPULATIONS | 8 |
| 9. | DATA CONVENTIONS FOR ANALYSIS | 8 |
| | 9.1 General Statistical Principles | 8 |
| | 9.2 Study Day | 9 |
| 10. | STATISTICAL EVALUATION | 9 |
| | 10.1 Subject Disposition | 9 |
| | 10.2 Protocol Deviation | 9 |
| | 10.3 Demographic and Baseline Characteristics | 9 |
| | 10.4 Study Drug Exposure and Compliance | 10 |
| | 10.5 Concomitant Medications | 10 |
| | 10.6 Medical History | 11 |
| | 10.7 Efficacy Endpoints | 11 |
| | 10.7.1 Primary Efficacy Endpoint | 11 |
| | 10.7.2 Secondary Efficacy Endpoints | 11 |
| | 10.8 Efficacy Analyses | 12 |
| | 10.8.1 Primary Efficacy Analysis | 12 |
| | 10.8.2 Secondary Efficacy Analysis | 13 |
| | 10.8.3Other Efficacy Analyses | 13 |
| | 10.9 Safety Analysis | 13 |
| | 10.9.1 Adverse Events | 13 |
| | 10.9.2 Application Site Reactions | 14 |
| | 10.9.3 Pregnancy Tests | 14 |

# Statistical Analysis Plan

| | 10.9.4Physical Examination | 14 |
|-----|--------------------------------------------------|----|
| | 10.9.5Vital Signs | 14 |
| 11. | CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES | 15 |
| 12. | HEADINGS | 15 |
| 13. | ARCHIVING AND RETENTION OF DOCUMENTS | 15 |
| 14. | OUTLINE OF PROPOSED TABLES, LISTINGS AND FIGURES | 15 |

# LIST OF SELECTED ABBREVIATIONS

| AD | Atopic Dermatitis |
|------|-------------------------------------------|
| ADR | Adverse Drug Reaction |
| AE | Adverse Event |
| BSA | Body Surface Area |
| CFR | Code of Federal Regulations |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| DMP | Data Management Plan |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practices |
| GLP | Good Laboratory Practices |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IGA | Investigator Global Assessment |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| ITT | Intention To Treat |
| LOCF | Last Observation Carried Forward |
| mITT | Modified Intention To Treat |
| OGD | Office of Generic Drugs |
| PI | Principal Investigator |
| PP | Per Protocol |
| SD | Standard Deviation |
| SAE | Serious Adverse Event |
| SAS | Statistical Analyzing System |
| SOP | Standard Operating Procedure |

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on protocol version 2.0 as issued on 14 October, 2016.

This document provides additional details concerning the statistical analyses outlined in the protocol and reflects any changes to the protocol from any amendments. This plan will not repeat all the definitions given in the protocol but will provide further details of the summaries and analyses planned therein.

#### 2. STUDY OBJECTIVES

#### **Primary Objective:**

• To establish the bioequivalence between test drug (Pimecrolimus Cream, 1%) and reference listed drug (Elidel® (pimecrolimus) Cream 1%) in the treatment of mild to moderate Atopic Dermatitis (AD), using the primary endpoint in the Per Protocol (PP) population, as detailed in FDA Draft Guidance on Pimecrolimus 1% Topical Cream dated March 2012.

#### **Additional Objectives:**

- To establish superiority of each active treatment over the placebo using the primary endpoint in the modified intent to treat (mITT) population and Last Observation Carried Forward (LOCF)
- To assess individual signs and symptoms of AD (i.e., erythema, induration/papulation, lichenification and pruritus) in each treatment group
- To compare the safety and tolerability between the test and reference drugs

#### 3. STUDY DESIGN

The study is a randomized, double blind, active and placebo controlled, prospective multicenter, comparative therapeutic equivalence study in which subjects with mild to moderate atopic dermatitis (AD) are randomized in a 1:1:1 allocation to test drug (Pimecrolimus Cream, 1%) or reference listed drug (RLD) (Elidel® (Pimecrolimus) Cream 1%) or placebo (vehicle cream). As per FDA recommendations, this study will be a bioequivalence study with a clinical endpoint in the treatment of mild to moderate AD comparing the test product versus the reference listed drug and vehicle control. A placebo control arm (vehicle of test product) is used to demonstrate that the test product and RLD are active and as a parameter to establish that the study is sufficiently sensitive to detect differences between products. The primary endpoint is the proportion of subjects with treatment success (a grade of clear or almost clear; a score of 0 or 1, within the

treatment area) based on the Investigator's Global Assessment (IGA) of Disease Severity at the end of treatment (study Day 15).

A total of 648 subjects will be included (216 in each active group and 216 in the placebo group). Subjects are non-immunocompromised males and females aged 8 years and above with mild to moderate atopic dermatitis who have failed to respond adequately to other topical prescription treatments, or when those treatments are not advisable.

The study duration for each subject would be up to 21 days, with a possible screening period of 14 days and a treatment period of 14 days. The study will include a total of 4 scheduled visits: screening visit (up to -14 days), baseline and randomization visit (day 1), interim visit (day  $8 \pm 3$  days), end of therapy visit (day  $15 \pm 3$  days).

Study kit numbers will be randomly assigned to one of the three treatment arms based on a randomization code list. The statistician will generate the randomization code list; a copy of this list will be shared with the IP handling team. Subjects fulfilling inclusion and exclusion criteria will receive study product from the next available sequential randomized kit which contains one of the three treatment arms. Each study product kit will contain three 100 gram tubes of study cream from the same randomized treatment arm. The kits will be packaged in a block size of 6. Each block will contain 2 kits of each treatment arm (Test: RLD: Placebo=2:2:2).

Efficacy assessments including Signs and Symptoms of Atopic Dermatitis will be scored per body region (head and neck; trunk; upper limbs; lower limbs) by the principal investigator or a qualified person delegated by the investigator at each visit. Pruritus will be assessed by questioning the subject or the subject's guardian regarding the intensity in the 24 hours prior to the visit for the overall condition. Overall Body Surface Area (BSA) Involvement with AD will be assessed and recorded by the investigator or delegate. Investigator's Global Assessment of Disease Severity Scoring will be scored for the investigator's (or delegate's) assessment of the subject's overall condition.

#### 4. HARDWARE AND SOFTWARE

Statistical analysis will be performed following Novella/TKL standard operating procedures and on the Novella computer network. All statistical analysis will be performed using SAS Version 9.3 with program code prepared specifically for the project by qualified Novella statisticians and SAS programmers.

The SAS programs will generate rich-text-formatted (RTF) output with the "RTF" extension using the SAS Output Delivery System (ODS). The summary tables and listings will be formatted using the Times New Roman 9-point font. The RTF output is included in report documents prepared with Microsoft Word and converted to PDF format without typographical change.

 *June 29, 2017* 

Datasets will be created and taken as input to validated SAS programs to generate the report-ready tables, listings, and figures. Each output display will show the names of the data sets and SAS program used to produce it.

#### 5. DATABASE CLOSURE

According to the Data Management Plan, after completion of all data review procedures, validation of the project database, and approval of the data review document by the study sponsor, the clinical database will be locked. Any change to the clinical database after this time will require written authorization, with explanation, by the Sponsor and the Biostatistician.

#### 6. SAMPLE SIZE DETERMINATION

The primary statistical analysis of interest is the proportion of subjects in the PP population with a clinical response of treatment success (at least an Investigator's Global Assessment of Clear or Almost Clear) at study Day 15. Considering the pivotal studies of the Reference Listed Drug, it is assumed that the active test and RLD will have approximate success rates at 21% and the vehicle cream will have an approximate success rate of 9%. A sample size of 184 subjects per group will provide at least 99% power to demonstrate bioequivalence (i.e., the 90% confidence interval (Yates' continuity -corrected) of the absolute difference between the test and reference composite success rates is within a defined equivalence range [-0.20, +0.20]). Assuming the conversion rate from mITT to PP will be about 90%, 205 subjects in each of the groups of the mITT population will provide at least 85% power to demonstrate superiority of active over placebo. Under the above assumptions, the overall global study power to demonstrate bioequivalence and superiority is estimated to be approximately 85%. To allow for about 5% of subjects who may drop out from the study or are otherwise non-evaluable, approximately 648 subjects will be enrolled (216 in each active group and 216 in the placebo group).

#### 7. HANDLING OF DROPOUTS AND MISSING DATA

For the analyses of the primary efficacy endpoint, subjects whose condition worsens and require alternate or supplemental therapy for the treatment of their AD during the study should be discontinued, included in the PP population analysis as treatment failures, and provided with effective treatment. Subjects discontinued early for other reasons should be excluded from the PP population, but included in the mITT population, using Last Observation Carried Forward (LOCF). For example, subjects who develop a skin infection in the treated area requiring treatment should be discontinued, excluded from the PP population, but included in the mITT population, using LOCF.

No missing imputations will be done for other non-primary efficacy endpoints or safety endpoints.

#### 8. ANALYSIS POPULATIONS

Four populations will be defined for analysis:

- <u>Safety population</u>: The safety population includes all randomized who received study product.
- <u>Modified ITT (mITT) population</u>: The mITT population includes all randomized subjects who met all inclusion/exclusion criteria, applied at least one dose of assigned product and returned for at least one post-baseline evaluation visit.
- Per Protocol (PP) population: The PP population includes all randomized subjects who met all inclusion/exclusion criteria, applied 75% to 125% of the assigned product for the specified duration of the study, did not miss the scheduled applications for more than 3 consecutive days, and completed the evaluation within the designated visit window (+/- 3 day) with no protocol violations that would affect the treatment evaluation. The subject's compliance will be verified by the use of subject diaries, and the protocol violations that would affect the treatment evaluation.

Subjects to be included in each population will be determined prior to the unblinding of the study.

The PP and mITT populations will be used for the analyses of efficacy endpoints. The PP population will be the primary population for the primary efficacy bioequivalence analysis. The mITT population will be used for the superiority analysis. The Safety population will be used for the analyses of safety endpoints.

All efficacy analyses will be conducted according to the randomized treatment assignment; all safety analyses will be conducted according to the treatment actually received.

#### 9. DATA CONVENTIONS FOR ANALYSIS

#### 9.1 General Statistical Principles

The purpose of the study is to evaluate the efficacy, safety and tolerability of Pimecrolimus Cream, 1% compared with reference listed drug Elidel® (pimecrolimus) Cream 1% as well as placebo vehicle cream in patients with AD using clinical endpoints. All statistical processing will be performed using the SAS system (Version 9.3).

All observed and derived variables (e.g., change from baseline, treatment success status) used in the summaries of analyses will be presented in by-subject listings. Descriptive statistics will be used to provide an overview of the efficacy and safety results. For categorical parameters, the number and percentage of subjects in each category will be presented. The denominator for percentage will be based on the number of subjects appropriate for the purpose of analysis. For continuous parameters, descriptive statistics will include number of observations, mean, standard deviation (SD), median, and range.

Small study centers with few subjects randomized will be pooled into analysis centers based on geographic locations. The pooling plan will be determined prior to the unblinding of the study.

Baseline value is defined as the last non-missing value prior to the first dose of study drug. Change from baseline is defined as the post-baseline value minus the baseline value.

No adjustments for multiple comparisons are planned. No interim analyses are planned.

#### 9.2 Study Day

Day 1 is defined as the date of first study drug administration or date of randomization for those subjects with missing date of first study drug administration. Study day is calculated relative to the date of Day 1.

#### 10. STATISTICAL EVALUATION

#### 10.1 Subject Disposition

The number and percentage of subjects who are screened, randomized, included in each analysis population, who complete the study, withdraw from the study (overall and by reason for withdrawal), and who are excluded from the PP population (overall and by reason for exclusion) will be summarized using frequencies and percentages by treatment group. The number of subjects who are enrolled and included in each study population will also be summarized for each study center.

A by-subject enrollment and disposition listing will be presented for all randomized subjects. Subjects who are screen failures and subjects who are not randomized will also be presented in a separate listing.

#### 10.2 Protocol Deviation

Protocol deviations will be presented in a by-subject listing, and summarized by treatment group in total per category.

#### **10.3** Demographic and Baseline Characteristics

Demographics and baseline characteristics will be summarized overall and by treatment for the Safety, mITT and PP populations. Statistical comparisons will be performed to detect any baseline differences between test and reference. Continuous variables will be compared using a two-sample t test; categorical variables will be compared using a Fisher's Exact test.

The following demographic and baseline variables will be included:

• Age with mean +/-SD and range

- Age group (<18 years,  $\ge18$  years)
- Sex N and %
- Ethnicity N and %
- Race N and %
- Body weight and height
- IGA
- Signs and symptoms:
  - o By body region: erythema, induration/papulation, and lichenification
  - o Overall: pruritus
- Percent Body Surface Area (BSA) (%)
- Application site reactions (dryness, burning/stinging, erosion, edema, and pain)
- Dermatological history, including:
  - o Dermatologic malignancy (Yes, No)
  - Reason for use of the study products

#### 10.4 Study Drug Exposure and Compliance

Assessments of study drug exposure and compliance will occur at Visit 3 (Day 8) and Visit 4 (Day 15) based on the treatment diary card. The following parameters will be summarized, by Day 8 and Day 15, for each treatment group for the mITT and PP populations:

- Number of days of exposure, defined as the date of last dose of study drug minus date of first dose of study drug plus 1
- Number of expected applications
- Number of applications
- Number of missed applications
- Percentage of compliance based on the investigator's review of subject diary, defined as the number of applications divided by the number of expected applications
- Subject compliance (Yes, No), defined as being 75%-125% in percent compliance

#### 10.5 Prior and Concomitant Medications

Prior (with stop dates prior to Day 1) and concomitant medications (ongoing or with stop dates on or after Day 1) for safety population will be provided separately in by-subject listings. If the medication is ongoing or the stop year is missing, the medication will be considered as received for the remainder of the study.

For the determination of prior vs concomitant medications, the following rules regarding the stop date will be applied:

• If only year was recorded, and it is before Baseline, it is a prior medication; if year is same or after Baseline, it is assumed to be a concomitant medication.

- If day is missing, but month and year are before Baseline, it is a prior medication; if month and year are the same as Baseline, it is assumed to be a concomitant medication; if month and year are after Baseline, it is a concomitant medication.
- If start date is after Baseline, it is a concomitant medication regardless.

Prior and concomitant medications will be summarized separately by treatment, WHO-DD Anatomical-Therapeutic-Chemical (ATC) classification and preferred term (PT).

#### **10.6** Medical History

Past and current medical conditions for all randomized subjects will be provided in a by-subject listing and summarized by treatment group. Dermatological history will be provided in a separate listing.

#### 10.7 Efficacy Endpoints

#### 10.7.1 Primary Efficacy Endpoint

The primary endpoint is the proportion of subjects with treatment success (i.e., a grade of clear or almost clear; a score of 0 or 1, within all treatment areas) at the end of treatment (Day 15) based on the IGA.

| IGA Score | Category |
|-----------|------------------|
| 0 | Clear |
| 1 | Almost Clear |
| 2 | Mild disease |
| 3 | Moderate disease |
| 4 | Severe disease |

#### 10.7.2 Secondary Efficacy Endpoints

Secondary efficacy endpoints will be the change from baseline to Day 15 in individual signs and symptoms of AD, including:

- Erythema (per body region, i.e., head and neck, trunk, upper limbs, and lower limbs)
- Induration/papulation (per body region)
- Lichenification (per body region)
- Pruritus (overall)

| Signs and Symptoms | Category |
|--------------------|----------|
| 0 | None |
| 1 | Mile |
| 2 | Moderate |

 *June 29, 2017* 

3 Severe

#### 10.8 Efficacy Analyses

#### 10.8.1 Primary Efficacy Analysis

#### **Equivalence Analysis**

Therapeutic equivalence of the test product (Pimecrolimus Cream, 1%) to the reference product (Elidel® (pimecrolimus) Cream 1%) will be evaluated using the PP population. If the 90% confidence interval (CI), with Yates' continuity correction of the test - reference difference for the primary endpoint (IGA success proportion) is contained within [-0.20, +0.20], then bioequivalence of the test product to the reference product will be considered to have been demonstrated.

The compound hypothesis to be tested is:

$$H_0$$
:  $P_T$  -  $P_R$  < -0.20 or  $P_T$  -  $P_R$  > 0.20

versus

$$H_A$$
:  $-0.20 \le P_T - P_R \le 0.20$ 

where  $P_T$  = success rate of test treatment and  $P_R$  = success rate of reference treatment.

Let

 $n_T$  = sample size of test treatment group Tn

 $cn_T$  = number of successes in test treatment group Tn

 $n_R$  = sample size of reference treatment group Rn

cn<sub>R</sub> = number of successes in reference treatment group Rn

$$P_T = cn_T / n_T$$
,  $P_R = cn_R / n_R$ , and  $se = (P_T (1 - P_T) / n_T + P_R (1 - P_R) / n_R) \frac{1}{2}$ .

The 90% CI for the difference in proportions between test and reference will be calculated as follows, using Yates' correction:

$$L = (P_T - P_R) - 1.645 \text{ se} - (1/n_T + 1/n_R)/2$$

$$U = (P_T - P_R) + 1.645 \text{ se} + (1/n_T + 1/n_R)/2$$

We reject  $H_0$  if  $L \ge -0.20$  and  $U \le 0.20$ . Rejection of the null hypothesis  $H_0$  supports the conclusion of equivalence of the two products.

#### **Superiority Analysis**

As a parameter for determining adequate study sensitivity, the test product and reference product will be compared to placebo with regard to the primary endpoint. Superiority of the test and

reference products against the placebo will be tested using Fisher's exact test in the mITT population with LOCF. The test and reference products should both be superior to placebo at the 5% significance level (p<0.05; two-sided) in order to claim adequate study sensitivity.

#### 10.8.2 Secondary Efficacy Analysis

The categorical change from baseline to Day 15 in individual signs and symptoms of AD per body region will be summarized using frequency counts and percentages.

#### 10.8.3 Other Efficacy Analyses

The overall BSA (%), along with the change from baseline values will be summarized using descriptive statistics by treatment group at each visit.

#### 10.9 Safety Analysis

All safety analyses will be based on the Safety Population according to the treatment received. .

#### 10.9.1 Adverse Events

AE terms will be coded using MedDRA dictionary. A treatment-emergent AE (TEAE) is defined as an AE that emerges during and after a certain period of treatment having been absent pretreatment, or worsen relative to the pre-treatment state. In case of partially recorded dates, similar rules as stated in section 10.5 regarding the start and stop date will be adopted. If relationship to treatment is missing, the event will be conservatively summarized as being related to study drug. If severity is missing, a separate category of missing severity will be included in the summary table, and no imputation of severity will be performed. Through the data cleaning process, all attempts will be made to avoid missing values for relationship and severity.

All AEs will be presented in a by-treatment and by-subject listing, detailing the verbatim term given by the investigator, the preferred term (PT), system organ class (SOC), onset date and time, end date and time, severity, outcome, relationship to study drug, action taken with study drug, other action taken, seriousness and criteria for seriousness. Serious AEs (SAEs) and TEAEs leading to study discontinuation will also be presented in a separate listing.

An overall summary of AEs will be presented by treatment and overall. The summary will include the frequency counts and percentages with:

- Any AE
- Any TEAE
- Any serious TEAE
- Any treatment-related TEAE, including definitely related, probably related, and possibly related

• Any TEAE leading to study drug discontinuation

Fisher's Exact test will also be performed to compare the incidence of the above between test and reference.

Summaries of the incidence of TEAEs will be displayed by treatment according to the following:

- All TEAEs by SOC in alphabetical order and PT in descending order of frequency (the combined frequency in the two active treatments)
- All TEAEs by SOC, PT, and maximum severity (mild, moderate, or severe)
- All TEAEs by SOC, PT, and maximum causality (not related, related) to the study drug

At each level of summarization, a subject will be counted once if he/she reported one or more events. The severity of TEAEs and relationship to study drug will be summarized in a similar manner. For summaries of relationship to study drug, a subject will be classified according to the closest relationship. For summaries of TEAE severity, a subject will be classified according to the highest severity.

#### **10.9.2** Application Site Reactions

Application site reactions including dryness, burning/stinging, erosion, edema, and pain, will be assessed based on Local Irritation Scale (LIS).

| Application site reactions | 0 | 1 | 2 | 3 |
|----------------------------|------|------|----------|--------|
| | None | Mild | Moderate | Severe |

Application site reaction scores will be summarized using frequency counts and percentages by visit for each treatment.

#### **10.9.3 Pregnancy Tests**

Urine pregnancy test results will be presented in a by-subject listing.

#### 10.9.4 Physical Examination

Abnormal physical examination results will be presented in a by-subject listing.

#### 10.9.5 Vital Signs

Vital sign parameters including pulse rate, blood pressure, and body temperature will be summarized using descriptive statistics at Baseline and Visit 4 (Day 15). By-subject listing will be presented.

#### 11. CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES

This SAP reflects the analysis plan outlined in the study protocol without significant change.

#### 12. HEADINGS

Each page of the analysis will show the sponsor's name, the investigational product, and the protocol number. Report tables will be embedded in the MS Word report document from SAS program output without change. The footer of each table will show the name of the SAS program module which generated it, the names of all data sets providing input data in the program and the date and time the table was generated.

### 13. ARCHIVING AND RETENTION OF DOCUMENTS

After finalization of the analysis, the following will be archived at Novella Clinical and/or with the study sponsor:

- SAP and any amendments
- All SAS code used in the project for statistical analysis, report tables generation, and analysis data set creation
- Tables, listings and figures as included in the clinical study report
- SAS study data tabulation model (SDTM) and analysis dataset model (ADaM) datasets.

#### 14. OUTLINE OF PROPOSED TABLES, LISTINGS AND FIGURES

# **Summary Tables**

| 14.1.1.1 | Subject Populations |
|---|---|
| 14.1.1.1.2 | Subject Populations by Site |
| 14.1.1.2.1 | Summary of Patient Discontinuation/Early Termination from the Study |
| 14.1.1.3 | Summary of Protocol Deviations; Safety Population |
| 14.1.2.1.1 | Summary of Subject Demographics; Safety Population |
| 14.1.2.1.2 | Summary of Subject Demographics; mITT Population |
| 14.1.2.1.3 | Summary of Subject Demographics; PP Population |
| 14.1.2.2.1 | Summary of Subject Baseline Characteristics; Safety Population |
| 14.1.2.2.2 | Summary of Subject Baseline Characteristics; mITT Population |
| 14.1.2.2.3 | Summary of Subject Baseline Characteristics; PP Population |
| 14.1.3 | Summary of Medical History; Safety Population |
| 14.1.4.1 | Summary of Prior Medications; Safety Population |
| 14.1.4.2 | Summary of Concomitant Medications; Safety Population |
| 14.1.5.1 | Summary of Study Medicaiton Exposure and Compliance; mITT Population |
| 14.1.5.2 | Summary of Study Medicaiton Exposure and Compliance; PP Population |
| 14.2.1 | Analysis of Primary Efficacy Oucome |
| 14.2.2.1.1 | Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Erythema by Body Region; PP Population |
| 14.2.2.1.2 | Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Erythema by Body Region; mITT Population |
| 14.2.2.2.1 | Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Induration/Papulation by Body Region; PP Population |
| 14.2.2.2.2 | Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Induration/Papulation by Body Region; mITT Population |
| 14.2.2.3.1 | Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Lichenification by Body Region; PP Population |
| 14.2.2.3.2 | Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Lichenification by Body Region; mITT Population |
| 14.2.2.4.1 | Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Overall Pruritus; PP Population |
| 14.2.2.4.2 | Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Overall Pruritus; mITT Population |
| 14.2.3.1 | Summary of Overall Body Surface Area by Visit; PP Population |
| 14.2.3.2 | Summary of Overall Body Surface Area by Visit; mITT Population |
| 14.3.1.1 | Overall Summary of Adverse Events; Safety Population |
| 14.3.1.2 | Summary of Treatment-emergent Adverse Events by System Organ Class and Preferred Term in Descending Frequency; Safety Population |
| 14.3.1.3 | Summary of Treatment-emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity; Safety Population |

| 14.3.1.4 | Summary of Treatment-emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Causality; Safety Population |
|---|---|
| 14.3.2 | Summary of Application Site Reactions; Safety Population |
| 14.3.3 | Summary of Vital Signs by Visit; Safety Population |

# Listing

| 16.1 | Subject Enrollment and Randomization; All Randomized Subjects |
|---|---|
| 16.2.1.1 | Screen Failures; All Screen Failure Subjects |
| 16.2.1.2 | Subject Disposition; All Randomized Subjects |
| 16.2.2 | Protocol Deviations |
| 16.2.3 | Population Inclusion; All Randomized Subjects |
| 16.2.4.1 | Demographics and Baseline Characteristics; All Randomized Subjects |
| 16.2.4.2.1 | Medical History; All Randomized Subjects |
| 16.2.4.2.2 | Dermatologial History and Diagnosis of AD; All Randomized Subjects |
| 16.2.4.3.1 | Prior Medications; All Randomized Subjects |
| 16.2.4.3.2 | Concomitant Medications; All Randomized Subjects |
| 16.2.5.1 | Study Drug Administration and Compliance; All Randomized Subjects |
| 16.2.5.2 | Subject Treatment Diary Card; All Randomized Subjects |
| 16.2.5.3 | Study Drug Accountability; All Randomized Subjects |
| 16.2.6.1 | Investigator's Global Assessment (IGA); All Randomized Subjects |
| 16.2.6.2 | Individual Signs and Symptoms of AD; All Randomized Subjects |
| 16.2.6.3 | Body Surface Area (BSA) Assessment; All Randomized Subjects |
| 16.2.7.1 | Adverse Events; All Randomized Subjects |
| 16.2.7.2 | Serious Adverse Events; All Randomized Subjects |
| 16.2.7.3 | Adverse Events Leading to Study Drug Discontinuation; All Randomized Subjects |
| 16.2.7.4 | Scoring of Local Application Site Reactions; All Randomized Subjects |
| 16.2.8.1 | Urine Pregnancy Test; All Randomized Subjects |
| 16.2.8.2 | Vital Signs; All Randomized Subjects |
| 16.2.8.3 | Physical Examination; Randomized Subjects with Abnormal Results |
| 16.2.9 | General Comments |


Table 14.1.1.1.1: Subject Populations

| | Pimecrolimus | Elidel® (Pimecrolimus) | | |
|---|---|---|---|---|
| | Cream, 1% | Cream, 1% | Placebo | Overall |
| Number of Subjects Enrolled | | | | XX |
| Number of Subjects Randomized | XX | XX | XX | XX |
| Total Safety Population, n(%) | XX | XX | XX | XX |
| Total Exclusion from Safety Population | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for Exclusion from Safety | | | | |
| No Record of First Dose | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total mITT Population, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total Exclusion from mITT Population | | | | |
| Reason for Exclusion from mITT | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| No Record of First Dose | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No Post-Treatment Data | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Etc. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <b>Total PP Population, n (%)</b> Total Exclusion from PP Population | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for Exclusion from PP | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Enrolled in Error | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-Up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-compliant (Dosing) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Outside Visit Window | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Randomized in Error | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Restricted Medication | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | | XX (XX.X) | XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Other | XX(XX.X) | $\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda)$ | $\Lambda\Lambda$ ( $\Lambda\Lambda.\Lambda$ ) | $\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda)$ |

Note: Denominator for percentages is the number of randomized subjects.

| DPT Laboratories |
|----------------------|
| Protocol CD-14-875 |
| Novella No. CT991616 |


DPT Laboratories Protocol No. CD-14-875 

Table 14.1.1.1.2: Subject Populations by Site

| Site Number | Principal Investigator and Location | Enrolled (N) | Included in Safety<br>Population (N) | Included in mITT Population (N) | Included in PP Population (N) |
|---|---|---|---|---|---|
| 01 | xxxxxxxx | XX | XX | XX | XX |
| 02 | XXXXXXXXX | XX | XX | XX | XX |


DPT Laboratories Protocol No. CD-14-875 

Table 14.1.1.2.1: Summary of Patient Discontinuation/Early Termination from the Study All Randomized Subjects

| | Pimecrolimus<br>Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus)<br>Cream, 1%<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| eason for Discontinuation, n (%) | | | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Worsening Signs/Symptoms | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Subject Withdrew Consent | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Investigator Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Study Medication Compliance <75% or >125% | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Drug is Unblinded | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Protocol Violation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pregnant | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Administrative Reasons | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Denominator for percentages is the number of randomized subjects.


Table 14.1.1.3: Summary of Protocol Deviations Safety Population

| | Pimecrolimus<br>Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus)<br>Cream, 1%<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Protocol Deviation Type, n (%) | | | | |
| Randomized in Error | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-Compliance | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow Up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Outside Visit Window | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Restricted Medication | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Etc. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Page X of Y

Table 14.1.2.1.X: Summary of Subject Demographics [Safety Population][mITT Population][PP Population]

| | | Pimecrolimus<br>Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus)<br>Cream, 1%<br>(N=XX) | Placebo<br>(N=XX) | P Value[1] |
|---|---|---|---|---|---|
| Age (years) | $\begin{aligned} \text{Mean} &\pm \text{SD} \\ \text{Minimum, Maximum} \end{aligned}$ | $XX.X \pm XX.XX$ $XX, XX$ | $XX.X \pm XX.XX$ $XX, XX$ | $XX.X \pm XX.XX$<br>XX, XX | 0.XXXX |
| Age Group, n (%) | <18 years<br>≥18 years | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | 0.XXXX |
| Gender, n (%) | Female<br>Male | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | 0.XXXX |
| Ethnicity, n (%) | Hispanic or Latino<br>Not Hispanic or Latino | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | 0.XXXX |
| Race, n (%) | White Black/African American Native Hawaiian/Other Pacific Islander Asian American Indian/Alaska Native Other [2] | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | 0.XXXX |

<sup>[1]</sup> Statistical comparisons will be performed to detect any baseline differences between test and reference. Continuous variables will be compared using a two-sample t test; categorical variables will be compared using a Fisher's Exact test.

<sup>[2]</sup> See listing 16.2.4.1 for other races.

Page X of Y

Table 14.1.2.2.X: Summary of Baseline Characteristics [Safety Population][mITT Population][PP Population]

| | Pimecrolimus<br>Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus)<br>Cream, 1%<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Weight (kg) | (2. 222) | (1, 12,2) | (* * | (1, 1212) |
| N | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| Height (cm) | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| Erythema by Body Region, n(%) | | | | |
| Head and Neck | | | | |
| 0 – None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| 3 – Severe | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| <continue for="" limbs,="" limbs<="" lower="" td="" trunk,="" upper=""><td>&gt;</td><td></td><td></td><td></td></continue> | > | | | |
| Induration/Papulation by Body Region, n(%) Head and Neck | | | | |
| 0 - None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc.></etc.> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| < Continue for Trunk, Upper Limbs, Lower Limbs | ` / | , | ` / | ` , |

Page X of Y

Table 14.1.2.2.X: Summary of Baseline Characteristics [Safety Population][mITT Population][PP Population]

| | Pimecrolimus Elidel® (Pimecrolimus) Cream, 1% Cream, 1% (N=XX) (N=XX) | | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| | (11 111) | (11 121) | (11 111) | (11 7414) |
| Lichenification by Body Region, n(%) Head and Neck | | | | |
| 0 – None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc.></etc.> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <continue for="" l<="" limbs,="" lower="" td="" trunk,="" upper=""><td>imbs&gt;</td><td>, ,</td><td>, ,</td><td>, ,</td></continue> | imbs> | , , | , , | , , |
| Overall Pruritus, n(%) | | | | |
| 0 – None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Percentage of BSA involvement (%) | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| IGA of Disease Severity, n(%) | | | | |
| 2 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[1]</sup> See listing 16.2.4.1 for other races.

Page X of Y

Table 14.1.2.2.X: Summary of Baseline Characteristics [Safety Population][mITT Population][PP Population]

| | Pimecrolimus | Elidel® (Pimecrolimus) | | |
|---|---|---|---|---|
| | Cream, 1% | Cream, 1% | Placebo | Overall |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Application Site Reaction - Dryness, n(%) | | | | |
| 0 – None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Application Site Reaction - Burning/Stinging, n(%) | | | | |
| 0 – None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 - Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Application Site Reaction - Erosion, n(%) | | | | |
| 0 – None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Application Site Reaction - Edema, n(%) | | | | |
| 0 – None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Novella No. CT991616

DPT Laboratories Protocol No. CD-14-875 Page X of Y

Table 14.1.2.2.X: Summary of Baseline Characteristics [Safety Population][mITT Population][PP Population]

| | Pimecrolimus | Elidel® (Pimecrolimus) | | |
|---|---|---|---|---|
| | Cream, 1% | Cream, 1% | Placebo | Overall |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Application site reaction - Pain, n(%) | | | | |
| 0 – None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Dermatologic Malignancy, n(%) | | | | |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for Use of this Product, n(%) | | | | |
| Failed to respond adequately to other topical | | | | |
| prescription treatments for AD | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other topical prescription treatments for AD not | | | | |
| advisable | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Page X of Y

Table 14.1.3: Summary of Medical History by System Organ Class and Preferred Term Safety Population

| System Organ Class<br>Preferred Term | Pimecrolimus<br>Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus)<br>Cream, 1%<br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|---|
| Subjects with any Medical History, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << System Organ Class >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << System Organ Class >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << System Organ Class >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Counts reflect numbers of subjects reporting one or more medical history that map to MedDRA (Version 19.1) system organ class or preferred term.

Page X of Y

Table 14.1.4.1: Summary of Prior Medications by Anatomical Therapeutic Chemical Class (ATC) and Preferred Term Safety Population

| | Pimecrolimus Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus) Cream 1%<br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|---|
| Subjects with any Prior Medication, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Anatomical Therapeutic Chemical Class >> | | | |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Anatomical Therapeutic Chemical Class >> | | | |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |

Note: Any medication with stop date prior to Day 1 is a "prior medication" and any medication with stop date on or after Day 1 is a "concomitant medication." Counts reflect number of subjects in each treatment group reporting one or more prior medication that map to the WHO Drug anatomical therapeutic chemical or preferred term. A subject may be counted once only in each row of the table.

Page X of Y

Table 14.1.4.2: Summary of Concomitant Medications by Anatomical Therapeutic Chemical Class (ATC) and Preferred Term Safety Population

| | Pimecrolimus Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus) Cream 1%<br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|---|
| Subjects with any Concomitant Medication, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Anatomical Therapeutic Chemical Class >> | | | |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Anatomical Therapeutic Chemical Class >> | | | |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX | XXXXX |

Note: Any medication with stop date prior to Day 1 is a "prior medication" and any medication with stop date on or after Day 1 is a "concomitant medication." Counts reflect number of subjects in each treatment group reporting one or more concomitant medication that map to the WHO Drug anatomical therapeutic chemical or preferred term. A subject may be counted once only in each row of the table.

Page X of Y

Table 14.1.5.X: Summary of Study Medication Exposure and Compliance [mITT Population][PP Population]

| | Pimecrolimus Cream, 1% (N=XX) | | ` | limus) Cream, 1%<br>XX) | Placebo<br>(N=XX) | |
|---|---|---|---|---|---|---|
| | By Visit 3<br>(Day 8) | By Visit 4<br>(Day 15) | By Visit 3<br>(Day 8) | By Visit 4<br>(Day 15) | By Visit 3<br>(Day 8) | By Visit 4<br>(Day 15) |
| Percentage of Compliance (%) [1] | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Subject 75%-125% Compliant, n (%) | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[1]</sup> Based on the investigator's review of subject diary, defined as the number of applications divided by the number of expected.

Page X of Y

Table 14.2.1: Analysis of Primary Efficacy Outcome IGA Success Rate on Day 15

| | Pimecrolimus<br>Cream, 1% | Elidel® (Pimecrolimus)<br>Cream, 1% | Placebo |
|---|---|---|---|
| P Population | | | |
| N | XX | XX | XX |
| IGA Success Rate, n/N (%) [1] | XX/XX (XX.XX) | XX/XX (XX.XX) | XX/XX (XX.XX) |
| 90% Confidence Interval Test – Reference [2] | XX.X | X, XX.XX | |
| nITT Population | | | |
| N | XX | XX | XX |
| IGA Success Rate, n/N (%) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| P-value, (Test or Reference) vs. Placebo [3] | 0.XXXX | 0.XXXX | |

<sup>[1]</sup> IGA success defined as achieving a grade of clear (0) or almost clear (1) on Day 15.

<sup>[2] 90%</sup> CI calculated with Yates' continuity correction. Equivalence of test to reference is considered to be demonstrated if the 90% CI is contained within [-0.20, +0.20].

<sup>[3]</sup> P-value calculated with Fisher's Exact Test.

Page X of Y

Table 14.2.2.1.X: Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis

Erythema by Body Region

[PP Population][mITT Population]

| | I | Pimecrolimus Cream, 1%<br>(N=XX) | | | Elidel | Elidel® (Pimecrolimus) Cream, 1% (N=XX) | | | | Placebo<br>(N=XX) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Head &<br>Neck | Trunk | Upper<br>Limbs | Lower<br>Limbs | Head &<br>Neck | Trunk | Upper<br>Limbs | Lower<br>Limbs | Head &<br>Neck | Trunk | Upper<br>Limbs | Lower<br>Limbs |
| Baseline | | | | | | | | | | | | |
| Observed Value, n (%) | | | | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 0 - None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 – Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 – Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 – Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 8 | | | | | | | | | | | | |
| Observed Value, n (%) | | | | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 0 - None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 – Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 – Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 – Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change From Baseline, | , n (%) | | | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 2 = Worsen by $2$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 = Worsen by $1$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 0 = No Change | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| -1 = Improve by 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| -2 = Improve by 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| -3 = Improve by 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Page X of Y

Table 14.2.2.1.X: Summary of Secondary Efficacy Outcome by Visit Individual Signs and Symptoms of Atopic Dermatitis

Erythema by Body Region

[PP Population][mITT Population]

| | I | Pimecrolimus Cream, 1%<br>(N=XX) | | | Elidel® (Pimecrolimus) Cream, 1% (N=XX) | | | | Placebo<br>(N=XX) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Head &<br>Neck | Trunk | Upper<br>Limbs | Lower<br>Limbs | Head &<br>Neck | Trunk | Upper<br>Limbs | Lower<br>Limbs | Head &<br>Neck | Trunk | Upper<br>Limbs | Lower<br>Limbs |
| Day 15 | | | | | | | | | | | | |
| Observed Value, n (% | <b>%</b> ) | | | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 0 - None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 – Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 – Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 – Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change From Baselin | ne, n (%) | | | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 2 = Worsen by $2$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 = Worsen by $1$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 0 = No Change | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| -1 = Improve by 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| -2 = Improve by 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| -3 = Improve by 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

#### <Repeat for >

Table 14.2.2.2.X: Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis

Induration/Papulation by Body Region

[PP Population][mITT Population]

Table 14.2.2.3.X: Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis

Lichenification by Body Region

[PP Population][mITT Population]

Page X of Y

# Table 14.2.2.4.X: Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Overall Pruritus [PP Population][mITT Population]

| · | Elidel® (Pimecrolimus) | | |
|---|---|---|---|
| | Pimecrolimus Cream, 1% | Cream, 1% | Placebo |
| | (N=XX) | (N=XX) | (N=XX) |
| Baseline | | | |
| Observed Value, n (%) | | | |
| N | XX | XX | XX |
| 0 - None | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Day 8 | | | |
| Observed Value, n (%) | | | |
| N | XX | XX | XX |
| 0 - None | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Change From Baseline, n (%) | | | |
| N | XX | XX | XX |
| 2 = Worsen by $2$ | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| 1 = Worsen by 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 0 = No Change | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| -1 = Improve by 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| -2 = Improve by 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| -3 = Improve by 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
Page X of Y

# Table 14.2.2.4.X: Summary of Secondary Efficacy Outcomes by Visit Individual Signs and Symptoms of Atopic Dermatitis Overall Pruritus [PP Population][mITT Population]

| | | Elidel® (Pimecrolimus) | |
|---|---|---|---|
| | Pimecrolimus Cream, 1% (N=XX) | Cream, 1% (N=XX) | Placebo<br>(N=XX) |
| Day 15 | | | |
| Observed Value, n (%) | | | |
| N | XX | XX | XX |
| 0 - None | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Change From Baseline, n (%) | | | |
| N | XX | XX | XX |
| 2 = Worsen by $2$ | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 = Worsen by $1$ | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 0 = No Change | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| -1 = Improve by 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| -2 = Improve by 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| -3 = Improve by 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Page X of Y

Table 14.2.3.X: Summary of Overall Body Surface Area by Visit [PP Population][mITT Population]

| | | Pimecrolimus Cream, 1% (N=XX) | | limus) Cream 1%<br>XX) | Plac<br>(N=) | |
|---|---|---|---|---|---|---|
| | · | Change from | | Change from | • | Change from |
| | Observed Value | Baseline | Observed Value | Baseline | Observed Value | Baseline |
| Baseline | | | | | | |
| N | XX | | XX | | XX | |
| Mean (SD) | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | |
| Median | XX.X | | XX.X | | XX.X | |
| Minimum, Maximum | XX.X, XX.X | | XX.X, XX.X | | XX.X, XX.X | |
| Day 8 | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Day 15 | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Page X of Y

Table 14.3.1.1: Overall Summary of Adverse Events All Randomized

| Description | Pimecrolimus<br>Cream, 1%<br>(N=XX) | Elidel®<br>(Pimecrolimus)<br>Cream 1%<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) | P Value[2] |
|---|---|---|---|---|---|
| Description | (N-AA) | (N-AA) | (N-AA) | (IV-AA) | r value[2] |
| Patients Randomized, n (%) | | | | | |
| Patients with at Least One Treatment-emergent AE (TEAE) [1] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Discontinued Study Drug Due to TEAE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| TEAEs Reported, n (%) | | | | | |
| Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Definite Related | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Probably Related | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Possibly Related | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Not Related | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Missing Relationship | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |
| Serious AE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | 0.XXXX |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA (Version XX). A subject may be counted once only in each row of the table.

<sup>[1]</sup> TEAEs are defined as AEs with an onset date on or after the date of the first applications of study medication.

<sup>[2]</sup> Fisher's Exact test will be performed to compare the incidence of the above between test and reference

DPT Laboratories
Page X of Y
Protocol No. CD-14-875

Table 14.3.1.2: Summary of Treatment-emergent Adverse Events by System Organ Class and Preferred Term in Descending Frequency Safety Population

| System Organ Class<br>Preferred Term | Pimecrolimus<br>Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus)<br>Cream 1%<br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|---|
| Subjects with any TEAE, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event System Organ Class >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| << Adverse Event System Organ Class >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX(XX.X) |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA (Version 19.1) system organ class or preferred term. A subject may be counted once only in each row of the table.

Generated on XX/XX/XX:XXXX by SMYTEAEPT / Uses: XXXX / Reference: Data Listings XXXX

<Programming Note: sort by SOC in alphabetical order and PT in descending order of the combined frequency in the two active treatments>

Page X of Y

Table 14.3.1.3: Summary of Treatment-emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Safety Population

| System Organ Class<br>Preferred Term | Severity | Pimecrolimus<br>Cream, 1%<br>(N=XX) | Elidel® (Pimecrolimus)<br>Cream 1%<br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|---|---|
| Treetrea Term | Severity | (11 7474) | (11 121) | (11, 121) |
| Subjects with any TEAE, n (%) | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event System Organ Class >> | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| • • | Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA (Version 19.1) system organ class or preferred term. A subject may be counted only once at the highest severity.

Page X of Y

Table 14.3.1.4: Summary of Treatment-emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Causality Safety Population

| | | Pimecrolimus | Elidel® (Pimecrolimus) | |
|---|---|---|---|---|
| System Organ Class | Causality | Cream, 1% | Cream 1% | Placebo |
| Preferred Term | Assessment[1] | (N=XX) | (N=XX) | (N=XX) |
| Subjects with any TEAE, n (%) | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Related | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| | Not Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event System Organ Class >> | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Not Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Not Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA (Version 19.1) system organ class or preferred term. A subject may be counted only once at the highest causality.

<sup>[1]</sup> Related includes definitely related, probably related, and possibly related events. If relationship to treatment is missing, the event will be conservatively summarized as being related to study drug

Page X of Y

Table 14.3.2: Summary of Application Site Reactions
Safety Population

| | Pimecrolimus Cream, 1%<br>(N=XX) | | | Elidel® (I | Pimecrolimus) (<br>(N=XX) | Cream 1% | Placebo<br>(N=XX) | | |
|---|---|---|---|---|---|---|---|---|---|
| | Baseline | Day 8 | Day 15 | Baseline | Day 8 | Day 15 | Baseline | Day 8 | Day 15 |
| Dryness, n(%) | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 0 - None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Stinging/burning, n(%) | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 0 - None | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Erosion, n(%) | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 0 - None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Page X of Y

Table 14.3.2: Summary of Application Site Reactions
Safety Population

| | Pimecrolimus Cream, 1%<br>(N=XX) | | | Elidel® ( | Pimecrolimus) C<br>(N=XX) | Cream 1% | Placebo<br>(N=XX) | | |
|---|---|---|---|---|---|---|---|---|---|
| | Baseline | Day 8 | Day 15 | Baseline | Day 8 | Day 15 | Baseline | Day 8 | Day 15 |
| Edema, n(%) | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 0 - None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pain, n(%) | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 0 - None | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Page X of Y

Table 14.3.3: Summary of Vital Signs by Visit Safety Population

| | Pimecrolimus Cream, 1%(N=XX) | | Elidel® (Pimecrolin<br>(N=X) | | Placebo<br>(N=XX) | |
|---|---|---|---|---|---|---|
| | Observed Value | Change from<br>Baseline | Observed Value | Change from<br>Baseline | Observed Value | Change from<br>Baseline |
| | Obscived value | Dascinic | Observed value | Dascinic | Observed value | Bascine |
| Body Temperature (°F) | | | | | | |
| Baseline | | | | | | |
| N | XX | | XX | | XX | |
| Mean (SD) | XX (XX.X) | | XX (XX.X) | | XX (XX.X) | |
| Median | XX (XX.X) | | XX (XX.X) | | XX (XX.X) | |
| Minimum, Maximum | XX, XX | | XX, XX | | XX, XX | |
| Day 15 | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Median | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

<sup>&</sup>lt; Continue for Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg), and Pulse Rate (bpm)>

Page X of Y

#### Data Listing 16.1: Subject Enrollment and Randomization All Randomized Subjects

| Subject<br>Number | Date and Time of Informed<br>Consent/Assent | Satisfy All<br>I/E Criteria? | Randomization<br>Date | Randomized<br>Kit Number | Randomized Treatment | Actual Treatment |
|---|---|---|---|---|---|---|
| | | N. T. 1 . W. | 1111111111111 | 3/3/3/3/ | P' 1' G 10/ | P' 1' G 10/ |
| XX-XXXX | YYYY-MM-DDTHH:MM | No: Inclusion XX | YYYY-MM-DD | XXXX | Pimecrolimus Cream, 1% | Pimecrolimus Cream, 1% |
| XX-XXXX | YYYY-MM-DDTHH:MM | Yes | YYYY-MM-DD | XXXX | Elidel® (Pimecrolimus) Cream 1% | Elidel® (Pimecrolimus) Cream 1% |
| XX-XXXX | YYYY-MM-DDTHH:MM | Yes | YYYY-MM-DD | XXXX | Placebo | Placebo |

Page X of Y

### Data Listing 16.2.1.1: Screen Failures All Screen Failure Subjects

| Subject<br>Number | Date and Time of Informed<br>Consent/Assent | Date of<br>Screening | Age<br>(Years) | Sex | Race | Ethnicity | Primary Reason for<br>Screen Failure |
|---|---|---|---|---|---|---|---|
| XX-XXXX | YYYY-MM-DDTHH:MM | YYYY-MM-DD | XX | X | XXXXXXXX | XXXXXXXX | I/E criteria not met: Inclusion 2 |
| XX-XXXX | YYYY-MM-DDTHH:MM | YYYY-MM-DD | XX | X | XXXXXXXX | XXXXXXXX | Other: XXXXXXX |
| XX-XXXX | YYYY-MM-DDTHH:MM | YYYY-MM-DD | XX | X | XXXXXXXX | XXXXXXXX | XXXXXXXXXX |
| XX-XXXX | YYYY-MM-DDTHH:MM | YYYY-MM-DD | XX | X | XXXXXXXX | XXXXXXXX | XXXXXXXXXX |
| XX-XXXX | YYYY-MM-DDTHH:MM | YYYY-MM-DD | XX | X | XXXXXXXX | XXXXXXXX | XXXXXXXXXX |

Page X of Y

## Data Listing 16.2.1.2: Subject Disposition All Randomized Subjects Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| | Date (Day) and Time of [1] | | | |
|---|---|---|---|---|
| First Treatment (Baseline) | Last Visit | Unblinding | Completion Status /<br>Discontinuation<br>Reason | Reason for Unblinding |
| | | 2 | | |
| YYYY-MM-DD (XX) | YYYY-MM-DD (XX)THH:MM | N/A | Completed | |
| YYYY-MM-DD(XX) | YYYY-MM-DD (XX)THH:MM | N/A | Lost to Follow-up | |
| YYYY-MM-DD(XX) | YYYY-MM-DD (XX)THH:MM | N/A | XXXXXXX | |
| YYYY-MM-DD (XX) | YYYY-MM-DD (XX)THH:MM | YYYY-MM-DD (XX) | XXXXXXX | XXXXXX |
| _ | YYYY-MM-DD (XX)<br>YYYY-MM-DD (XX)<br>YYYY-MM-DD (XX) | First Treatment (Baseline) Last Visit YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM | First Treatment (Baseline) Last Visit Unblinding YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM N/A YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM N/A YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM N/A | First Treatment (Baseline) Last Visit Unblinding Completion Status / Discontinuation Reason YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM N/A Completed YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM N/A Lost to Follow-up YYYY-MM-DD (XX) YYYY-MM-DD (XX)THH:MM N/A XXXXXXX |

<sup>[1]</sup> Day is date minus Baseline date plus 1.


DPT Laboratories Protocol No. CD-14-875 Page X of Y

### Data Listing 16.2.2: Protocol Deviations Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | Deviations/Violations<br>Done by | Category | Date of Deviation | Reason(s) for Deviation/Violations |
|---|---|---|---|---|
| XX-XXXX | Investigator | Major | YYYY-MM-DD | XXXXXXXX |
| XX-XXXX | Subject | Minor | YYYY-MM-DD | XXXXXXXX |

Page X of Y

## Data Listing 16.2.3: Population Inclusion All Randomized Subjects Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject | Safety | mITT | PP | | |
|---|---|---|---|---|---|
| Number | Population | Population | Population | Reason for Exclusion from mITT Population | Reason for Exclusion from PP Population |
| XX-XXXX | Yes | Yes | No | NA | Not compliant with the treatment regimen |
| | | | | | No Day 15 IGA evaluation within the designated |
| XX-XXXX | Yes | Yes | No | NA | visit window |
| XX-XXXX | Yes | No | No | Did not return for post-baseline visit | |
| XX-XXXX | Yes | No | No | Not meeting all inclusion/exclusion criteria | |

Page X of Y

### Data Listing 16.2.4.1: Demographics and Baseline Characteristics All Randomized Subjects

Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject | | | | ] | BSA Involvemen | t | | |
|---|---|---|---|---|---|---|---|---|
| Number | Age (Years) | Sex | Ethnicity | Race | (%) | IGA | Weight (kg) | Height (cm) |
| XX-XXXX | XX.X | X | XXXXXXXX | XXXXXX | XX.X | 2 - Mild | XX.X | XX.X |
| XX-XXXX | XX.X | X | XXXXX | Other: XXXXX | XX.X | 3 – Moderate | XX.X | XX.X |

Note: BSA = Body Surface Area; IGA = Investigator's Global Assessment

Page X of Y

## Data Listing 16.2.4.2.1: Medical History All Randomized Subjects Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | Diagnosis and/or Procedure | System Organ Class | Preferred Term | Onset Date | Resolution Date |
|---|---|---|---|---|---|
| XX-XXXX | XXXXXXXX | XXXXXXXX | XXXXXXX | XXXX-XX-XX | XXXX-XX-XX |
| | XXXXXXXX | XXXXXXXX | XXXXXXXX | XXXX-XX-XX | Ongoing |
| | XXXXXXXX | XXXXXXX | XXXXXXX | XXXX-XX-XX | XXXX-XX-XX |
| XX-XXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXX-XX-XX | XXXX-XX-XX |
| XX-XXXX | XXXXXXXX | XXXXXXXX | XXXXXXXX | XXXX-XX-XX | XXXX-XX-XX |

Page X of Y

### Data Listing 16.2.4.2.2: Dermatologial History and Diagnosis of AD All Randomized Subjects

Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject | Dermatologic | Reason for Use of | Dermatological | Hani | ifin and Rajka Criteria |
|---|---|---|---|---|---|
| Number | malignancy? | Study Products[1] | | Major | Minor |
| X- | Y | Inadequate prior | XXXXXX | XXXXXX | XXXXXX |
| XXX | _ | response | XXXXXXXXX | XXXXXXX | XXXXXXXXXXXXXX |
| | | - | | XXXXXXXXXXXXXXXXX | XXXXXXX |
| Х- | N | Cannot use other | XXXXXX | XXXXXX | XXXXXX |
| XXX | 11 | topicals | | XXXXXXXX | XXXXXXXXXXXXXX |
| | | | | XXXXXXXXXXXXXXXX | XXXXXXX |

<sup>[1]</sup> Inadequate prior response = failed to respond adequately to other topical prescription treatments for AD; Cannot use other topicals = it is not advisable for the subject to use other topical prescription treatments?

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX

<Programming note: concatenate and present all recorded reasons for use of study proudcts, derm exam results, and major and minor criteria >


DPT Laboratories Protocol No. CD-14-875 Page X of Y

### Data Listing 16.2.4.3.1: Prior Medications All Randomized Subjects

Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | WHO Preferred Term<br>(Verbatim Term) /<br>ATC Classification | Indication | Dosage / Units | Frequency / Route | Start Date (Day) – Stop Date (Day) [1] |
|---|---|---|---|---|---|
| | XXXXXXXX<br>(XXXXXXXX)/ | | | | |
| XX-XXXX | XXXXXXXX<br>XXXXXXXX<br>(XXXXXXXX)/ | Adverse Event | XXXX / XXXX | XXXX / XXXX | YYYY-MM-DD(X)- YYYY-MM-DD(X) |
| | XXXXXXXX | Medical History | XXXX / XXXX | XXXX / XXXX | YYYY-MM-DD(X)- Ongoing |

[1] Day is date of visit minus Baseline/Day 1 date plus 1.


DPT Laboratories Protocol No. CD-14-875 Page X of Y

## Data Listing 16.2.4.3.2: Concomitant Medications All Randomized Subjects Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | WHO Preferred Term<br>(Verbatim Term) /<br>ATC Classification | Indication | MH/AE SOC/<br>PT | Dosage / Units | Frequency / Route | Start Date (Day) – Stop Date (Day) [1] |
|---|---|---|---|---|---|---|
| XX-XXXX | XXXXXXXX<br>(XXXXXXXX) /<br>XXXXXXXX<br>XXXXXXXX | Adverse Event | XXXXXX | XXXX / XXXX | XXXX / XXXX | YYYY-MM-DD(X)- YYYY-MM-DD(X) |
| | (XXXXXXXX)/<br>XXXXXXXX | Medical History | XXXX | XXXX / XXXX | XXXX / XXXX | YYYY-MM-DD(X)- Ongoing |

<sup>[1]</sup> Day is date of visit minus Baseline/Day 1 date plus 1.

Page X of Y

## Data Listing 16.2.5.1: Study Drug Administration and Compliance All Randomized Subjects Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | Visit | Date of First Dose<br>Administration(AM/PM)/<br>Date of Last Dose<br>Administration(AM/PM) | Study Drug<br>Administration<br>Stopped? | Reason Stopped | Date (Day) of Decision[1] | Number of<br>Recorded<br>Doses | Number of<br>Expected<br>Doses | Percentage of<br>Compliance<br>(%) |
|---|---|---|---|---|---|---|---|---|
| | | YYYY-MM-DD (AM)/ | | | | | | |
| XX-XXXX | Day 8 | YYYY-MM-DD(XX) | No | NA | NA | XX | XX | XX.X |
| | | YYYY-MM-DD (PM)/ | | | | | | |
| | Day 15 | YYYY-MM-DD (XX) | Yes | XXXXXXX | YYYY-MM-DD(XX) | XX | XX | XX.X |
| | | YYYY-MM-DD (AM)/ | | | | | | |
| XX-XXXX | Day 8 | YYYY-MM-DD(XX) | No | NA | NA | XX | XX | XX.X |
| | | YYYY-MM-DD (PM)/ | | | | | | |
| | Day 15 | YYYY-MM-DD (XX) | Yes | XXXXXXX | YYYY-MM-DD(XX) | XX | XX | XX.X |

<sup>[1]</sup> Day is date of visit minus Baseline date plus 1.

Page X of Y

### Data Listing 16.2.5.2: Subject Treatment Diary Card All Randomized Subjects

Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject | Medication Application | Medicatio | on Applied | | Comments or Feeling of Discomfort Due to |
|---|---|---|---|---|---|
| Number | Date (Day)[1] | AM | PM | Reason if Medication not Applied | Medication |
| XX-XXXX | YYYY-MM-DD(1) | Y | N | XXXXXXX | XXXXX |
| | YYYY-MM-DD (XX) | Y | Y | NA | NA |

[1] Day is date minus Baseline date plus 1.

Page X of Y

### Data Listing 16.2.5.3: Study Drug Accountability All Randomized Subjects

Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| | | | <b>Used Drug Tubes</b> | | Unused/Pai | rtially Used l | Drug Tubes | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Visit | Date (Day)[1] | Collected? | Number<br>Used | Collected? | Number<br>Partially<br>Used | Number<br>unused | All Tubes Returned?/<br>Reason if Not | Study Drug Re-<br>dispensed?/<br>Reason if Not | Dispensing Date |
| | | YYYY-MM-DD | | | | | | No/ | Yes/ | |
| XX-XXXX | Day 8 | (XX) | Y | X | N | 0 | 0 | XXXXXXX | NA | YYYY-MM-DD |
| | | YYYY-MM-DD | | | | | | Yes/ | No/ | |
| | Day 15 | (XX) | N | 0 | Y | X | X | NA | XXXXX | NA |

[1] Day is date minus Baseline date plus 1.

Page X of Y

### Data Listing 16.2.6.1: Investigator's Global Assessment (IGA) All Randomized Subjects

Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| | | | | | Obser | rved | LOC | = | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Visit | Date (Day) [1] | Was IGA<br>Performed? | Reason if not<br>Performed | Overall IGA[2] | Change from Baseline[3] | Overall IGA | Change from<br>Baseline | IGA Success<br>on Day 15 |
| XX-XXXX | Screening | YYYY-MM-DD (XX) | Yes | NA | 2 – Mild | - | - | - | - |
| | Baseline/Day 1 | YYYY-MM-DD (XX) | Yes | NA | 2 - Mild | - | - | - | - |
| | Day 8 | YYYY-MM-DD (XX) | Yes | NA | 1 – Almost Clear | -1 | - | - | - |
| | Day 15 | $YYYY\text{-}MM\text{-}DD\left( XX\right)$ | Yes | NA | XXXXXX | X | XXXXXX | X | Y |

Note: Baseline is the last available measurement prior to first application of study medication. LOCF=Last Observation Carried Forward

<sup>[1]</sup> Day is date of visit minus Baseline date plus 1.

<sup>[2]</sup> Based on a 5-point scale of 0 (Clear) to 4 (Severe Disease).

<sup>[3]</sup> Indication: 2 = Worsen by 2 Points; 1 = Worsen by 1 Point; 0 = No Change; -1 = Improve by 1 Point; -2 = Improve by 2 Points; -3 = Improve by 3 Points

<sup>[4]</sup> LOCF results only present at Day 15

Page X of Y

## Data Listing 16.2.6.2: Individual Signs and Symptoms of AD All Randomized Subjects Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| | | | | Er | ythema | | ] | Indurati | on/Papulat | tion | | Liche | enification | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | • | Head & | | Upper | Lower | Head & | | Upper | Lower | Head & | | Upper | Lower | Overall |
| Number | Visit | Date (Day) [1] | Neck | Trunk | Limbs | Limbs | Neck | Trunk | Limbs | Limbs | Neck | Trunk | Limbs | Limbs | Pruritus |
| XX- | Screening | YYYY-MM-DD | | | | | | | | | | | | | |
| XXXX | | (XX) | 1 | X | X | X | X | X | X | X | X | X | X | X | X |
| | Baseline/Day | YYYY-MM-DD | | | | | | | | | | | | | |
| | 1 | (XX) | 3 | X | X | X | X | X | X | X | X | X | X | X | X |
| | Day 8 | YYYY-MM-DD | | | | | | | | | | | | | |
| | | (XX) | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | Day 15 | YYYY-MM-DD | | | | | | | | | | | | | |
| | - | (XX) | X | X | X | X | X | X | X | X | X | X | X | X | X |

Note: 0=None, 1=Mild, 2=Moderate, 3= Severe [1] Day is date minus Baseline date plus 1.

Page X of Y

#### Data Listing 16.2.6.3: Body Surface Area (BSA) Assessment All Randomized Subjects

Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | Visit | Date (Day) [1] | Was BSA Assessment Performed? | Reason if not<br>Performed | Percentage of BSA<br>Involvement (%) | Change from Baseline[2] |
|---|---|---|---|---|---|---|
| XX-XXXX | Screening | YYYY-MM-DD(XX) | Yes | NA | XX.X | - |
| | Baseline/Day 1 | YYYY-MM-DD (XX) | Yes | NA | XX.X | - |
| | Day 8 | YYYY-MM-DD (XX) | No | XXXXXX | XX.X | XX.X |
| | Day 15 | YYYY-MM-DD (XX) | Yes | NA | XX.X | XX.X |

Note: Baseline is the last available measurement prior to first application of study medication.

<sup>[1]</sup> Day is date of visit minus Baseline date plus 1.

<sup>[2]</sup> Calculated as post-Baseline minus Baseline.

Page X of Y

#### Data Listing 16.2.7.1: Adverse Events All Randomized Subjects Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | MedDRA SOC Term/<br>MedDRA Preferred Term /<br>(Verbatim Term) | SAE? SAE Criteria | Treatment-emergent? [1]<br>Onset Date (Day) –<br>End Date (Day) [2] | Outcome | Severity | Causality<br>Assessment | Action Taken /<br>Other Action<br>Taken |
|---|---|---|---|---|---|---|---|
| XX-XXXX | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | Yes: XXXXX | Yes /<br>YYYY-MM-DD (XX) –<br>YYYY-MM-DD (XX) | XXXXXXX | Mild | Definitely Related | XXXXXXXX /<br>XXXXXXXX |
| | XXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | No | No /<br>YYYY-MM-DD (XX) –<br>YYYY-MM-DD (XX) | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX /<br>XXXXXXXX |
| XX-XXXX | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | No | XXX /<br>YYYY-MM-DD (XX) –<br>YYYY-MM-DD (XX) | XXXXXXX | XXXXXXXX | XXXXXXX | XXXXXXXX /<br>XXXXXXXX |

Generated on XX/XX/XX:XXXX by LSTAE / Uses: AE

<sup>[1]</sup> Treatment-emergent AEs (TEAEs) are defined as AEs with an onset date on or after the first application of study medication. [2] Day is date minus Baseline/Day 1 date plus 1.

Page X of Y

#### Data Listing 16.2.7.2: Serious Adverse Events All Randomized Subjects Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | MedDRA SOC Term/<br>MedDRA Preferred Term /<br>(Verbatim Term) / | SAE Criteria | Treatment-emergent? [1]<br>Onset Date (Day) –<br>End Date (Day) [2] | Outcome | Severity | Causality Assessment | Action Taken /<br>Other Action Taken |
|---|---|---|---|---|---|---|---|
| XX-XXXX | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | XXXXX | Yes /<br>YYYY-MM-DD (XX) –<br>YYYY-MM-DD (XX) | XXXXXXXX | Mild | Definitely Related | XXXXXXXX /<br>XXXXXXXX |
| | XXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | XXXXX | No /<br>YYYY-MM-DD (XX) –<br>YYYY-MM-DD (XX) | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX /<br>XXXXXXXX |
| XX-XXXX | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | XXXXX | XXX /<br>YYYY-MM-DD (XX) –<br>YYYY-MM-DD (XX) | XXXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX /<br>XXXXXXXX |

Generated on XX/XX/XX:XXXX by LSTAE / Uses: AE

<sup>[1]</sup> Treatment-emergent AEs (TEAEs) are defined as AEs with an onset date on or after the first application of study medication. [2] Day is date minus Baseline/Day 1 date plus 1.

Page X of Y

### Data Listing 16.2.7.3: Adverse Events Leading to Study Drug Discontinuation All Randomized Subjects

Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | MedDRA SOC Term/<br>MedDRA Preferred Term /<br>(Verbatim Term) / | SAE? SAE<br>Criteria | Treatment-emergent? [1]<br>Onset Date (Day) –<br>End Date (Day) [2] | Outcome | Severity | Causality Assessment | Other Action Taken |
|---|---|---|---|---|---|---|---|
| XX-XXXX | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | Yes: XXXXX | $\begin{array}{l} Yes \ / \\ YYYY-MM-DD \ (XX) - \\ YYYY-MM-DD \ (XX) \end{array}$ | XXXXXXXX | Mild | Definitely Related | XXXXXXX |
| | XXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | No | No /<br>YYYY-MM-DD (XX) –<br>YYYY-MM-DD (XX) | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| XX-XXXX | XXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | No | XXX /<br>YYYY-MM-DD (XX) –<br>YYYY-MM-DD (XX) | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |

<sup>[1]</sup> Treatment-emergent AEs (TEAEs) are defined as AEs with an onset date on or after the first application of study medication.

<sup>[2]</sup> Day is date minus Baseline/Day 1 date plus 1.

Page X of Y

### Data Listing 16.2.7.4: Scoring of Local Application Site Reactions All Randomized Subjects

Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject | | | Was the Scoring | Reason not | | Stinging/ | | | _ |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Date (Day) [1] | Performed? | Performed | Dryness | Burning | Erosion | Edema | Pain |
| XX-XXXX | Screening | YYYY-MM-DD(XX) | Yes | NA | 1 – Mild | XXXX | XXXX | XXXX | XXXX |
| | Baseline/Day 1 | YYYY-MM-DD (XX) | Yes | NA | XXXX | XXXX | XXXX | XXXX | XXXX |
| | Day 8 | YYYY-MM-DD (XX) | Yes | NA | XXXX | XXXX | XXXX | XXXX | XXXX |
| | Day 15 | YYYY-MM-DD (XX) | Yes | NA | XXXX | XXXX | XXXX | XXXX | XXXX |

[1] Day is date of visit minus Baseline date plus 1.


DPT Laboratories Protocol No. CD-14-875 Page X of Y

#### 16.2.8.1: Urine Pregnancy Test All Randomized Female Subjects

Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | Childbearing Potential | Visit | Date of Test (Day)[1] | Result |
|---|---|---|---|---|
| | | | . •//. | |
| XX-XXXX | Abstinence | Baseline/Day 1 | YYYY-MM-DD (XX) | Negative |
| | | Day 15 | YYYY-MM-DD (XX) | Negative |
| XX-XXXX | XXXXXXX | Baseline/Day 1 | YYYY-MM-DD (XX) | Negative |
| | | Day 15 | YYYY-MM-DD (XX) | Negative |

[1]Day is date minus Baseline/Day 1 date plus 1.

Page X of Y

## Data Listing 16.2.8.2: Vital Signs All Randomized Subjects Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| | | | | | | Body Temp | | SBI<br>(mml | | DBI<br>(mmF | | Pulse Rate | e (bpm) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Visit | Date (Day) [1] | Assessment Performed? | Height (cm) | Weight<br>(kg) | Observed | CFBL | Observed | CFBL | Observed | CFBL | Observed | CFBL |
| XX-XXXX | Screening | YYYY-MM-DD (XX) | Y | XX.X | XX.X | XX.X | | xx.x | | xx.x | | xx.x | |
| | Baseline/Day 1 | YYYY-MM-DD (XX) | N:XXXX | XX.X | XX.X | xx.x (CS) | | XX.X | | XX.X | | XX.X | |
| | Day 8 | YYYY-MM-DD (XX) | Y | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Day 15 | YYYY-MM-DD (XX) | Y | XX.X | xx.x | XX.X | XX.X | xx.x (CS) | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX-XXXX | Screening | YYYY-MM-DD (XX) | Y | XX.X | xx.x | XX.X | | XX.X | | XX.X | | xx.x | |
| | Baseline/Day 1 | YYYY-MM-DD (XX) | Y | XX.X | XX.X | XX.X | | XX.X | | XX.X | | XX.X | |
| | Day 8 | YYYY-MM-DD (XX) | Y | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Day 15 | YYYY-MM-DD (XX) | Y | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Note: CS=Clinically Significant; SBP=Systolic blood pressure; DBP=Diastolic blood pressure; CFBL= change from baseline [1] Day is date of visit minus Baseline date plus 1.

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX

cprogramming note: include CS in bold for CS observations >

Page X of Y

### Data Listing 16.2.8.3: Physical Examination Randomized Subjects with Abnormal Results

Actual Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject<br>Number | Visit | Date (Day) [1] | Organ/System | Comment |
|---|---|---|---|---|
| XX-XXXX | Screening | YYYY-MM-DD (XX) | Head | XXXXXXXXX |
| | | | Eyes | XXXXX |
| | Baseline/Day 1 | YYYY-MM-DD(XX) | Eyes | XXXXXXXXX |
| XX-XXXX | XXXX | YYYY-MM-DD (XX) | NA | XXXXX |
| | XXXX | YYYY-MM-DD (XX) | Head | XXXXX |

<sup>[1]</sup> Day is date of visit minus Baseline date plus 1.

Page X of Y

### 16.2.9: General Comments Randomized Treatment: [Pimecrolimus Cream, 1%][Elidel® (Pimecrolimus) Cream 1%][Placebo]

| Subject | | |
|---------|--------------|-----------------------------------------|
| Number | Reference | Comment |
| XX-XXXX | eCRF Page XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | eCRF Page XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XX-XXXX | eCRF Page XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | eCRF Page XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |



Status: Completed

Ivelisse.Rivera@novellaclinical.com

IP Address: 65.205.190.115

Sent: 6/29/2017 7:53:08 AM

Sent: 6/29/2017 7:56:46 AM

**Timestamp** 

**Certificate Of Completion** 

Envelope Id: 64D898E58F71424D8C9E3689337E9547

Subject: Please DocuSign: DPT CD-14-875 SAP Final.pdf

Source Envelope:

Document Pages: 68 Signatures: 3 **Envelope Originator:** Initials: 0 Supplemental Document Pages: 0 Ivelisse Rivera

Certificate Pages: 5

AutoNav: Enabled Payments: 0 1700 Perimeter Park Drive Morrisville, NC 27560

Envelopeld Stamping: Disabled

Time Zone: (UTC-08:00) Pacific Time (US &

Canada)

**Record Tracking** 

Status: Original Holder: Ivelisse Rivera Location: DocuSign

6/29/2017 7:49:51 AM Ivelisse.Rivera@novellaclinical.com

Signature Signer Events

Carol Udell Carol Udell Carol.Udell@novellaclinical.com

(Required)

Viewed: 6/29/2017 7:56:12 AM Security Level: Email, Account Authentication Signed: 6/29/2017 7:56:42 AM

Signature ID:

CE741CD0-FE97-41EC-A29C-B39E84B183BB

Using IP Address: 65.205.190.115

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 6/29/2017 6:05:59 AM

ID: 23a67abb-661c-48d7-a3b0-5cd8fbe94ff5

Katrin Beckmann

Katrin Beckmann katrin.beckmann@mylan.com Viewed: 6/30/2017 1:51:15 AM

Security Level: Email, Account Authentication Signed: 6/30/2017 2:15:07 AM

Signature ID:

(Required)

57B7C204-8BC8-4782-AF97-02CCDE55D6D2

Using IP Address: 129.35.202.236

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 6/30/2017 1:51:15 AM

ID: 9581a9a6-b595-476f-993b-ccbfcdd15ba0

| Signer Events | Signature | Timestamp |
|---|---|---|
| Kathleen Ocasio<br>Kathleen.Ocasio@dptlabs.com | Kathleen Ocasio | Sent: 6/30/2017 2:15:11 AM<br>Resent: 6/30/2017 5:34:01 AM |
| Security Level: Email, Account Authentication (Required) | Signature ID:<br>FFE08E0F-E0E3-411F-89EF-D4D82881E090<br>Using IP Address: 67.86.42.245 | Resent: 6/30/2017 5:59:52 AM Resent: 7/6/2017 8:05:31 AM Viewed: 6/30/2017 6:37:50 AM Signed: 7/7/2017 6:38:00 AM |
| Electronic Record and Signature Disclosure: | With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document | d |

Accepted: 6/30/2017 6:37:50 AM ID: c4951be6-83ed-40c1-adfb-38d49d6344c2

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Jonathan Prado<br>Jonathan.Prado1@novellaclinical.com<br>Security Level: Email, Account Authentication | COPIED | Sent: 7/7/2017 6:38:05 AM<br>Viewed: 7/7/2017 6:39:43 AM |

(Required)

Electronic Record and Signature Disclosure: Not Offered via DocuSign

| Notary Events | Signature | Timestamp |
|---------------------------------|------------------|---------------------|
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 7/7/2017 6:38:05 AM |
| Certified Delivered | Security Checked | 7/7/2017 6:38:05 AM |
| Signing Complete | Security Checked | 7/7/2017 6:38:05 AM |
| Completed | Security Checked | 7/7/2017 6:38:05 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature | Disclosure | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Novella Clinical DocuSign Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### **How to contact Novella Clinical DocuSign Part 11:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: ngliatis@novellaclinical.com

#### To advise Novella Clinical DocuSign Part 11 of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at ngliatis@novellaclinical.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

### To request paper copies from Novella Clinical DocuSign Part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to ngliatis@novellaclinical.com and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

### To withdraw your consent with Novella Clinical DocuSign Part 11

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to ngliatis@novellaclinical.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| required hard ware and sortware | |
|---|---|
| Operating Systems: | Windows2000? or WindowsXP? |
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy<br>Server must enable HTTP 1.1 settings via<br>proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Novella Clinical DocuSign Part 11 as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Novella Clinical DocuSign Part 11 during the course of my relationship with you.